CLINICAL TRIAL: NCT05916287
Title: HÉRITABILITÉ FAMILIALE, INTERACTIONS GÈNE-GÈNE ET GÈNE-ENVIRONNEMENT DANS LE DOMAINE DES MALADIES CARDIOVASCULAIRES ET RENALES. Cinquième Visite de la Cohorte STANISLAS
Brief Title: FAMILY INHERITANCE, GENE-GENE AND GENE-ENVIRONMENT INTERACTIONS IN THE FIELD OF CARDIOVASCULAR AND RENAL DISEASES. Fifth Visit of the STANISLAS Cohort
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr. Nicolas GIRERD, Coordinating doctor, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020PI129; 2021-A00449-32 (Other: ANSM)
Record Dates: First submitted 2023-06-02; First posted 2023-06-23 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Diseases; Cohort Studies; Genotype; Risk Factors; Nutrition
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Blood Specimen Collection; Eating; Ambulatory Care Facilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volonteer (Experimental)
  Interventions: Biological: Blood and urine samples; Genetic: Blood samples; Other: Cardiovascular assessment; Behavioral: Dietary intake; Other: Anthropometric parameters; Other: Hemodynamic parameters; Behavioral: Assessment of compliance with antihypertensive treatments for treated participants; Other: Ambulatory 24 hours measurment of blood pressure; Biological: 24 hours urinary collection; Other: General questionnaires; Other: Women specific questionnaire; Behavioral: Women specific questionnaire; Diagnostic Test: NYHA dyspnea questionnaire; Behavioral: Anxiety questionnaire; Behavioral: Epworth Sleepiness Scale; Other: A questionnaire on the "perception of the management of cardiovascular risk factors"; Behavioral: A questionnaire on eating behaviors; Behavioral: A questionnaire on eating habits to determine consumer profiles; Dietary Supplement: A questionnaire on food supplements use; Other: SARS-CoV-2 Infection Questionnaire; Other: Instantaneous expired air analysis; Biological: Capillary sampling

INTERVENTIONS:
Biological: Blood and urine samples — Blood and urine samples
Genetic: Blood samples — Blood samples
Other: Cardiovascular assessment — Echocardiography, Lung ultrasound, pulse wave velocity, carotid stiffness and thickness, Central and peripheral blood pressure, carotid pulse pressure, abdominal aorta ultrasound, jugular vein ultrasound, liver elastography (Optional).
Behavioral: Dietary intake — Food frequency questionnaires, ''Dutch eating behaviour questionnaire'' and dietary supplement questionnaire
Other: Anthropometric parameters — Measurement of height, weight, abdominal circumference, hip circumference, arm circumference
Other: Hemodynamic parameters — Systolic pressure index measurement
Other: Hemodynamic parameters — Heart rate measurements, blood pressure measurements, orthostatic BP measurements
Other: Hemodynamic parameters — Blood pressure measurements by "unattended BP" monitor over 5 min
Other: Hemodynamic parameters — Electrocardiogram
Behavioral: Assessment of compliance with antihypertensive treatments for treated participants — EVALOBS scale and compliance questionnaire
Other: Ambulatory 24 hours measurment of blood pressure — For the first 100 patients willing to participate
Biological: 24 hours urinary collection — For the first 100 patients willing to participate. For biobank constitution and measurement of microalbuminuria, creatininuria, osmolarity, natriuresis, kaliuresis, urea, proteinuria and urine dipstick
Other: General questionnaires — Collection of socio-demographic data such as age, level of education, profession, household income, smoking status, physical activity, perception of health, prematurity, height and weight at birth, family and personal history especially cardiovascular (history of stroke, myocardial infarction, heart failure, current pathologies, drugs, tobacco...)
Other: Women specific questionnaire — Women specific questionnaire
Behavioral: Women specific questionnaire — Women specific questionnaire
Diagnostic Test: NYHA dyspnea questionnaire — Determination of NYHA class.
Behavioral: Anxiety questionnaire — Assessment of anxiety
Behavioral: Epworth Sleepiness Scale — sleep quality assessment
Other: A questionnaire on the "perception of the management of cardiovascular risk factors" — Patient's evaluation of cardiovascular risk factors by the health system
Behavioral: A questionnaire on eating behaviors — Assessment of eating behaviors
Behavioral: A questionnaire on eating habits to determine consumer profiles — Assessement of eating habit to create a consumer profile
Dietary Supplement: A questionnaire on food supplements use — Evaluation od food supplements intake
Other: SARS-CoV-2 Infection Questionnaire — SARS-CoV-2 Infection Questionnaire
Other: Instantaneous expired air analysis — Carbon monoxyde analysis in expired air
Biological: Capillary sampling — Capillary sampling for pollutant analysis (Optional)

SUMMARY:
The Stanislas Cohort is a monocentric familial longitudinal cohort originally comprised of 1006 families consisting of two parents and at least two biological children and deemed healthy, recruited in 1993-1995 at the Centre for Preventive Medicine of Nancy. This cohort was established with the primary objective of investigating gene-gene and gene-environment interactions in the field of cardiovascular diseases. The 5th visit of the STANISLAS Cohort will allow a better evaluation of the cardiovascular ageing of the population and the transition toward cardiovascular or renal diseases in relation with their genetic profile and environment.

DETAILED DESCRIPTION:
The main objective of the STANISLAS cohort is to identify the factors associated with cardiovascular aging (assessed through the study of the degradation of morphological and functional parameters of the heart and vascular systems).

Data (clinical, biological, morphological, genetic and lifestyle) from previous visits (the first having been initiated in the mid-1990s) will be considered as exposure and / or adjustment variables.

The exposure variables of interest will be:

* The components of metabolic syndrome (MS),
* Genetic determinants, through an approach of family segregation and candidate genes,
* Multi-omic biomarkers analyzed from the biological collection of the first assessments of the cohort
* Food intake, nutrition and eating behavior

The secondary objectives are

* Identify the factors associated with a degradation of renal parameters (renal function and proteinuria).
* Identify the factors associated with a degradation of metabolic parameters.
* To assess the association between SARS-CoV-2 infection (questionnaire and serological approach) and cardiovascular and renal parameters
* Identify factors associated with the occurrence of clinical cardiovascular events.
* Association between Covid 19 events and general disabling symptoms
* Complete the cohort's biological collection for future biomarker assays related to previous objectives

ELIGIBILITY:
Inclusion Criteria:

* aged over 18
* Person who participated in the Stanislas Cohort
* Person affiliated to a social security scheme or beneficiary of such a scheme
* Person having received complete information on the organization of the research and having signed an informed consent

Exclusion Criteria:

* Persons deprived of their liberty by a judicial or administrative decision, persons undergoing psychiatric treatment under Articles L. 3212-1 and L. 3213-1
* Person referred to in Articles L. 1121-5, L. 1121-7 and L1121-8 of the Public Health Code:

  * Pregnant woman, parturient or nursing mother
  * Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
  * Person of full age unable to express consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2027-07-13 (Estimated); Study Completion 2027-07-13 (Estimated)

PRIMARY OUTCOMES:
Indexed left ventricular mass measured by echocardiography | Baseline
Left ventricular volume measured by echocardiography | Baseline
Tissue doppler imaging e' wave measured by echocardiography | Baseline
Ratio E/e' measured by echocardiography | Baseline
Left atrial volume measured by echocardiography | Baseline
Pulmonary congestion evaluated by lung ultrasound | Baseline
Pulse wave velocity measured by Sphygmocor and Complior Analyse | Baseline
Carotid intima media thickness measured by echotracking | Baseline
Central blood pressure | Baseline

SECONDARY OUTCOMES:
Estimation of the glomerular filtration rate (CKD-EPI formula) | Baseline
  Composite endpoint of degradation of renal function (With outcome 11)
Proteinuria (on sample) | Baseline
  Composite endpoint of degradation of renal function (With outcome 10)
Blood glucose | Baseline
  Composite endpoint of degradation of metabolic parameters (With outcome 13 and 14)
Change in HbA1C | Baseline
  Composite endpoint of degradation of metabolic parameters (With outcome 12 and 14)
Change in lipid parameters (LDL and HDL cholesterol) | Baseline
  Composite endpoint of degradation of metabolic parameters (With outcome 12 and 13)
Occurrence of the following clinical CV events: Hospitalization for HF, HF not requiring hospitalization, Atrial fibrillation, Acute coronary syndrome, Coronary artery disease, Hypertension (requiring introduction of drug treatment), Stroke | Baseline
General symptoms persisting beyond 8 weeks after SARS-CoV-2 infection such as: disabling asthenia, disabling dyspnea, cardiothoracic signs, arthromyalgia, neurocognitive disorders or anosmia | Baseline
Results of future relevant biomarker assays | Baseline
  Biomarkers on the cardiovascular field, measured on biological collection and dependant on the progress of knowledge and technology

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Girerd, MD, PhD, Principal Investigator — Centre d'Investigation Clinique 1433 module Plurithématique - CHRU Nancy
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, Lorraine, France